CLINICAL TRIAL: NCT04534582
Title: A Randomised, Parallel, Single-Dose, Subcutaneous Injection, Phase I Clinical Study Of HLX14 Versus Prolia® (Denosumab) In Chinese Healthy Adult Male Subjects For Comparison In Pharmacokinetic Characteristics, Safety, And Immunogenicity
Brief Title: Pharmacokinetic, Safety and Immunogenicity Phase I Study of HLX14 Versus Prolia® in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX14-001
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-03

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part I: open label Part II: masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part I: HLX14 group (Experimental): Part I: HLX14 are given subcutaneous injection at a single dose of 60 mg.
  Interventions: Drug: HLX14
- Part I: EU-Prolia® group (Active Comparator): Part I: EU-Prolia® are given subcutaneous injection at a single dose of 60 mg.
  Interventions: Drug: EU-Prolia®
- Part II: HLX14 group (Experimental): Part II: HLX14 are given subcutaneous injection at a single dose of 60 mg.
  Interventions: Drug: HLX14
- Part II: EU-Prolia® group (Active Comparator): Part II: EU-Prolia® are given subcutaneous injection at a single dose of 60 mg.
  Interventions: Drug: EU-Prolia®
- Part II: US-Prolia® group (Active Comparator): Part II: US-Prolia® are given subcutaneous injection at a single dose of 60 mg.
  Interventions: Drug: US-Prolia®
- Part II: CN-Prolia® group (Active Comparator): Part II: CN-Prolia® are given subcutaneous injection at a single dose of 60 mg.
  Interventions: Drug: CN-Prolia®

INTERVENTIONS:
Drug: HLX14 — healthy volunteers receive HLX14 (60mg) once
  Arms: Part I: HLX14 group; Part II: HLX14 group
Drug: EU-Prolia® — healthy volunteers receive EU-Prolia® (60mg) once
  Arms: Part I: EU-Prolia® group; Part II: EU-Prolia® group
Drug: US-Prolia® — healthy volunteers receive US-Prolia® (60mg) once
  Arms: Part II: US-Prolia® group
Drug: CN-Prolia® — healthy volunteers receive CN-Prolia® (60mg) once
  Arms: Part II: CN-Prolia® group

SUMMARY:
Part I of the study： This is a randomised, single-dose, subcutaneous injection, parallel study designed to compare the PK of HLX14 and EU-sourced Prolia® in healthy Chinese adult male subjects, and to assess the safety, tolerability, and immunogenicity of these 2 drugs.

Part II of the study： This is a randomised, double-blind, four-arm, single-dose, subcutaneous injection, parallel-controlled study to evaluate the PK, PD, safety, tolerability, and immunogenicity between-group following a single subcutaneous injection of HLX14 or US, EU, CN-sourced Prolia®.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged> 28 and ≤ 65 years;
2. Body weight ≥ 50 kg, body mass index (BMI) = body weight (kg)/body height2 (m2), BMI ≥ 19 and ≤ 26 kg/m2;
3. With no disease history, or with abnormal prior medical history which has no effect on the trial as judged by the physician;
4. Normal or abnormal without clinical significance in physical examination, vital signs, ECG, chest imaging, clinical laboratory test, etc.;
5. Before the trial, sign the informed consent form (ICF) and have a full understanding of trial content, process, and possible adverse events (AEs); be able to complete the study as per protocol requirements.

Exclusion Criteria:

1. With a history of allergy to study drugs, calcium, and/or vitamin D, or with a history of allergy to drugs or others not suitable for participating in this study as judged by the investigators;
2. With the following clinically significant diseases (including but not limited to digestive system, kidney diseases, liver diseases, nervous diseases, blood system, endocrine system, tumor, respiratory system, immune diseases, mental diseases, cardiovascular and cerebrovascular diseases, or any condition that may affect bone metabolism);
3. With a history of upper respiratory tract infection and other acute infections within 2 weeks prior to screening;
4. Occurred or suffering from osteomyelitis or ONJ (Osteonecrosis of the jaw) previously.

   The dental or jaw disease that is active, requiring oral surgery; or dental or oral surgery wounds have not healed; or planned for invasive dental surgery during the study.
5. Occurrence of fracture or bone-related surgery within 6 months prior to screening;
6. With rash, scar, tattoo, etc. at administration site that may affect drug absorption;
7. Blood donation or massive blood loss (> 450 mL) within 3 months prior to screening;
8. Use of any prescription drugs, over-the-counter (OTC) drugs, vitamin products, or traditional Chinese medicines within 28 days prior to screening;
9. Participation in any drug clinical trials and use of any investigational/comparator drugs within 3 months prior to screening;
10. Administration of the following drugs affecting bone metabolism:

    1. Administration history of denosumab or its biosimilar products, romosozumab or its biosimilar products, cathepsin K inhibitors, diphosphonates, fluorides, or stronitum;
    2. Administration of the following within 12 months before screening: parathyroid hormone or its derivatives, hormone replacement therapy (HRT), selective estrogen receptor modulators (SERM), tibolone, anabolic steroids, testosterone, androgen, and gonadotropin-releasing hormone agonists (GnRH-a);
    3. Administration of any prescription drug or OTC drug within 6 months or 10 half-lives of drug elimination (whichever is the longer) before screening that may have impact on the objectives of the study at the discretion of the investigator, including but not limited to heparin, warfarin, anticonvulsants (excluding benzodiazepine), systemic ketoconazole, adrenocorticotropic hormone (ACTH), cinacalcet, aluminum, lithium, protease inhibitors (PI), methotrexate (MTX), calcitonin, calcitriol, diuretics, and glucocorticoids for oral administration or injection (daily administration of ≥ 5 mg prednisone or equivalent drugs for more than 10 days);
11. Use of any biological products (excluding vaccine) or monoclonal antibodies within 6 months prior to screening;
12. Vaccination within 1 month prior to screening;
13. With a history of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, 25 mL of spirit, or 100 mL of wine), or positive for alcohol breath test;
14. With a history of substance abuse or drug abuse, or positive for drug screen;
15. Positive for tobacco screen;
16. With significant changes in physical activity within 6 months prior to screening, or not agree to abstain from strenuous physical exercise during the trial;
17. Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody (TPPA);
18. Abnormal serum calcium level (beyond the laboratory reference range) during the screening;
19. Ear temperature > 37.5 °C during the screening period; and/or sitting systolic blood pressure (SBP) > 140 mmHg or < 90 mmHg, and/or diastolic blood pressure (DBP) > 90 mmHg or < 50 mmHg; and/or pulse rate > 100 beats/min or < 50 beats/min during the screening.
20. Clinically significant abnormal ECG or QTcF > 450 ms during screening, or with a prior history of clinically significant abnormal ECG;
21. Unwilling to take adequate contraceptive measures during the study.
22. Subjects who, in the opinion of the investigators, are not eligible to participate in this study.

Ages: 28 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | from 0 to day 274
  Area under the serum concentration-time curve from time 0 to the last concentration-quantifiable time t of denosumab
Cmax | from 0 to day 274
  Maximum serum concentration following administration of denosumab
AUC0-inf | from 0 to day 274
  Area under the serum concentration-time curve from time 0 to infinity

SECONDARY OUTCOMES:
Tmax | from 0 to day 274
  Time to reach maximum serum concentration following administration
CL/F | from 0 to day 274
  Total clearance
λz | from 0 to day 274
  Apparent terminal elimination rate constant
t1/2 | from 0 to day 274
  Elimination half life
Vd/F | from 0 to day 274
  Apparent volume of distribution
%AUCex | from 0 to day 274
  Area extrapolated from time to infinity as a percentage of total AUC0-inf
MRT | from 0 to day 274
  Mean residence time
AUC0-28d and AUC0-112d | from 0 to day 112
  Area under the drug concentration-time curve from day 0 to day 28 (4 weeks) and from day 0 to day 112 (16 weeks)
AUEC0-t | from 0 to day 274
  Area under the effect-time curve from time zero to last time of quantifiable concentration of serum CTX1
Imin | from 0 to day 274
  Minimum observed concentration of serum CTX1
Imax | from 0 to day 274
  Maximum percent inhibition of serum CTX1
Tmin | from 0 to day 274
  Time to reach Imin of serum CTX1

OTHER OUTCOMES:
AEs and SAEs | from 0 to day 274
  Adverse events and serious adverse events
Physical examination | from 0 to day 274
Vital signs | from 0 to day 274
Injection site reactions | from 0 to day 274
Laboratory tests (haematology, serum chemistry, and urinalysis) | from 0 to day 274
12-lead ECG | from 0 to day 274
ADA and NAb | from 0 to day 274
  Positive rate of anti-drug antibody, including neutralising antibody

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li N, Chu N, Zhu L, Wu X, Wei Q, Wang J, Hu X, Yu H, Wang Q, Yuan W, Huang K, Zhang J. Pharmacokinetics, pharmacodynamics, safety, and immunogenicity of HLX14 versus reference denosumab in healthy males: A randomized phase I study. Clin Transl Sci. 2024 Dec;17(12):e70089. doi: 10.1111/cts.70089. PMID 39700054
- [Result] American Society for Clinical Pharmacology and Therapeutics. Clin Pharmacol Ther. 2022 Mar;111 Suppl 1:S5-S80. doi: 10.1002/cpt.2521. No abstract available. PMID 35132630